CLINICAL TRIAL: NCT02556294
Title: Fostering Resilience to Psychosocial and HIV Risk in Indian MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The National Institute for Research in Tuberculosis (Unknown); Indian Council of Medical Research (Other Government); Sahodaran (Unknown); The Humsafar Trust (Unknown); Fenway Community Health (Other)
Responsible Party: Principal Investigator, Steven A. Safren, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH100627-01A1 (NIH); R01MH100627-01A1 (NIH)
Record Dates: First submitted 2015-04-23; First posted 2015-09-22 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: HIV Infection; Sexual Behavior; Health Behavior
Keywords: HIV risk behavior
MeSH Terms: conditions — HIV Infections; Sexual Behavior; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-acceptance behavioral intervention (Experimental): The intervention will consist of individual and 4 group counseling sessions and 6 individual counseling sessions. The individual sessions are focused on specific individualized risk reduction plans, whereas the group sessions are focused on increasing self-acceptance and reducing HIV risk. Additionally, participants in this arm will receive HIV and STI counseling and testing.
  Interventions: Behavioral: Self-acceptance based intervention; Behavioral: HIV/STI counseling and testing
- Comparison/Control (Other): The comparison group will receive HIV and STI counseling and testing.
  Interventions: Behavioral: HIV/STI counseling and testing

INTERVENTIONS:
Behavioral: Self-acceptance based intervention — The intervention will consist of HIV/STI counseling and testing as well as individual counseling sessions and group sessions. The primary focus of the group sessions are to help foster self-acceptance by the support from the group, as well as learn skills to reduce distress and HIV risk. The primary purpose of the individual sessions is to help develop and implement an individualized plan for HIV risk reduction, and, as needed and available, linkage to other services.
  Arms: Self-acceptance behavioral intervention
Behavioral: HIV/STI counseling and testing — The counseling component is standard of care in India and will focus on HIV/STI risk and how to minimize risk. This is followed by biological testing for HIV and STIs.

SUMMARY:
India has the world's third largest HIV epidemic and men who have sex with men (MSM) are an identified high risk group. MSM in India face unique psychosocial stress underlying the context of HIV risk. To maximize the potential impact of an HIV prevention intervention, the purpose of this study is to test, in a two-arm randomized controlled efficacy trial, a behavioral intervention that addresses both psychosocial / contextual stress and reducing participant's risk for HIV.

DETAILED DESCRIPTION:
India has the world's third largest HIV epidemic, and MSM in India have an estimated seroprevalence of 14.7%. Many HIV prevention efforts for MSM in India are limited to condom distribution and HIV education, with no existing efficacy trials of HIV prevention interventions and therefore no evidenced based HIV prevention interventions this population. MSM in India are hidden, stigmatized, and face considerable psychosocial stressors, including pressure to marry, which potentially increases the risk for HIV transmission to their wives.

This proposal is the culmination of our ongoing, successful > 10-year community based research collaboration with two NGOs dedicated to HIV prevention among MSM, Sahodaran (Chennai) and The Humsafar Trust (Mumbai), and investigators from the India Council of Medical Research (ICMR), National Institute for Research in Tuberculosis (NIRT) in Chennai. Our work, including extensive community advisory input, has identified self-acceptance as a key resilience variable that protects against both HIV risk and psychosocial distress. A field test and pilot randomized controlled trial of our behavioral intervention that addresses both HIV risk and self-acceptance showed high participant acceptability and feasibility of study procedures, and success reducing HIV sexual risk behavior.

The current study is a two-arm randomized controlled trial to reduce HIV, STI and sexual transmission risk compared to HIV/STI counseling and testing alone.

ELIGIBILITY:
Inclusion Criteria - One of the following must be true:

* Participant has had anal sex with 4 or more male partners (protected or unprotected) in the past 4 months.
* Participant has had condomless anal sex with a man who was HIV unknown or serodiscordant in the past 4 months.
* Participant has a history of transactional sex activity in the past 4 months.
* Participant has been given a diagnosis of an STI in the past 4 months.

Exclusion Criteria:

* Participant does not identify as male
* Younger than 18
* Is unable to understand or consent to the procedures
* Is deemed by the local PI or study staff to be engaging in deception about the inclusion/exclusion criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Changes in frequency of condomless sex | 4 month visit, 8 month visit, 12, month visit
  Self-reported insertive or receptive anal sex without the use of a condom.
Number of incident STIs from Baseline | 12 month visit
  Chlamydia, gonorrhea, syphilis, and HIV

SECONDARY OUTCOMES:
Changes in Psychosocial Mediators | Measured at baseline, 4, 8, 12 month visits
  Items will be used to measure potential psychosocial mediators (e.g. self-acceptance questionnaire, distress questionnaire) at each major visit.
Cost-effectiveness of intervention | 12 months
  To assess the incremental cost-effectiveness of the experimental versus the comparison condition.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Safren, PhD, Principal Investigator — University of Miami; Matthew J Mimiaga, ScD, MPH, Principal Investigator — Brown University; Conall M O'Cleirigh, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- India (2):
  - The National Institute for Research in Tuberculosis, Chennai
  - The Humsafar Trust, Mumbai

REFERENCES:
- [Derived] Safren SA, Thomas B, Biello KB, Mayer KH, Rawat S, Dange A, Bedoya CA, Menon S, Anand V, Balu V, O'Cleirigh C, Klasko-Foster L, Baruah D, Swaminathan S, Mimiaga MJ. Strengthening resilience to reduce HIV risk in Indian MSM: a multicity, randomised, clinical efficacy trial. Lancet Glob Health. 2021 Apr;9(4):e446-e455. doi: 10.1016/S2214-109X(20)30547-7. PMID 33740407
- [Derived] Mimiaga MJ, Thomas B, Mayer KH, Regenauer KS, Dange A, Andres Bedoya C, Rawat S, Balu V, O'Cleirigh C, Biello KB, Anand V, Swaminathan S, Safren SA. A randomized clinical efficacy trial of a psychosocial intervention to strengthen self-acceptance and reduce HIV risk for MSM in India: study protocol. BMC Public Health. 2018 Jul 18;18(1):890. doi: 10.1186/s12889-018-5838-2. PMID 30021566